CLINICAL TRIAL: NCT07340671
Title: Evaluating the Efficacy of the 1726nm Laser for the Treatment of Facial Papules in Frontal Fibrosing Alopecia (FFA)
Brief Title: Facial Papules in Frontal Fibrosing Alopecia (FFA)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Cutera Inc. (Industry)
Responsible Party: Principal Investigator, Ariel Eva Eber, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250543
Record Dates: First submitted 2025-12-01; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Frontal Fibrosing Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 1726 nm Laser Treatment Group (Experimental): Participants will be in this group for up to approximately 30 weeks and complete up to 5 visits
  Interventions: Device: Cutera® 1726 nm laser system

INTERVENTIONS:
Device: Cutera® 1726 nm laser system — Participants will receive 3 laser treatments at 4 (±1) week intervals and will be followed at approximately at 12 (± 2) weeks post treatment completion onsite.
  Other Names: Cutera®; AviClear®

SUMMARY:
The objective is to evaluate the safety and efficacy of the Cutera 1726 nm laser system (also referred to as AviClear) for the treatment of facial papules in frontal fibrosing alopecia (FFA).

ELIGIBILITY:
Inclusion Criteria:

* Female or Male
* Fitzpatrick Skin Types I-VI
* At least 18 years of age
* Has clinically diagnosed FFA with facial papules.
* Subject must be able to read, speak, and understand English or Spanish and sign the Informed Consent Form.
* Willing and able to adhere to the treatment and follow-up schedule and pre/post-treatment care instructions.
* No contraindication to laser therapy.
* Willing to have photographs taken of the treatment area and agree to the use of photographs for presentation, educational or marketing purposes.
* Agree to not undergo any other procedure(s) or add any new treatment modalities in the treatment area during the study.
* Willing to use investigator approved skincare topicals and follow investigator approved skincare regimen for the duration of the study.

Exclusion Criteria:

* Prior treatment to the target area during participation in a clinical trial of another device or drug within 1 month (30 days) prior to study participation.
* Prior treatment to the target area within 3 months of study participating including chemical peel, dermabrassion, microneedling, radiofrequency treatment, laser or light-based procedures, cryodestruction or chemodestruction, intralesional steroids, photodynamic therapy, or acne surgery.
* Prior injection of botulinum toxin in the target area within 3 months of study participation and for the duration of the study.
* Systemic use of retinoid, such as isotretinoin, within 3 months of study participation.
* Still healing from another treatment in the target area according to investigator's discretion.
* History of malignant tumors in the target area.
* Pregnant and/or breastfeeding or planning to become pregnant during the study.
* Suffering from diagnosed immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
* History of diagnosed connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the target area, unless treatment is conducted following a prophylactic regimen.
* History of radiation to the target area, currently undergoing treatment for skin cancer in the target area, or undergoing systemic chemotherapy for the treatment of cancer.
* History of diagnosed pigmentary disorders (including vitiligo) in the target area.
* Excessively tanned in the treatment area or unable/unlikely to refrain from tanning in the target area during the study.
* History of keloids or hypertrophic scarring.
* Prisoners
* As per the Investigator's discretion, any physical, mental or medical condition which might make it unsafe for the subject to participate in this study, might interfere with patient's participation in the full study protocol, or might interfere with the diagnosis or assessment of facial papules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in lesion size (papule diameter in mm) measured by dermatoscope and ultrasound | Baseline (Pretreatment), immediately after each treatment session, and at 12 week follow up
  Lesion size will be assessed using dermatoscope and ultrasound imaging. Measurements will be recorded in millimeters (mm) and compared to baseline values to evaluate treatment response.

SECONDARY OUTCOMES:
Change in lesion count measured by physical examination | Baseline (Pretreatment) immediately after each treatment, and at 12 week follow up
  Lesions will be counted manually during physical examination at each time point. Counts will be compared to baseline to assess treatment response
Change in lesion depth measured by optical coherence tomography (OCT) and/or ultrasound | Baseline (Pretreatment) immediately after each treatment, and at 12 week follow up
  Using optical coherence tomography (OCT) and/or ultrasound to measure subsurface changes, including lesion depth and size. Measurements will be compared to baseline to evaluate treatment response.
Change in appearance of facial papules assessed by standardized global photography | Baseline (Pretreatment), immediately after each treatment, and at 12 week follow up
  Facial papule appearance will be documented using standardized global photographs at each time point. Images will be evaluated for visual changes compared to baseline.
Change in Physician Global Assessment (PGA) score (9-point ordinal scale) | Baseline (Pretreatment) and 12 week follow up
  A board-certified physician will evaluate overall lesion severity using a standardized 9-point ordinal scale. Scores range from 0-8, with higher scores indicate greater severity. Scores at follow-up will be compared to baseline to assess treatment response.
Blinded dermatologist evaluation | Up to 30 weeks
  Before and after photos will be provided to three blinded dermatologists. Dermatologists will be asked to identify the correct before and after photos. Correct identification greater than or equal to 80% percent of the time is considered statistically significant.
Patient's self-assessment (PSA) scale | At baseline and through the completion of the study, approximate time of 30 weeks
  The Patient Self-Assessment (PSA) is a standardized patient-reported outcome measure of subjective improvement. Patients will rate their improvement using a 5-point Likert scale (1 = no improvement, 5 = significant improvement).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No